CLINICAL TRIAL: NCT00701376
Title: Long Term Hepatic Effects of Gastric Bypass Surgery
Brief Title: Hepatic Effects of Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-877
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Liver Diseases
Keywords: Gastric Bypass surgery; Hepatic disease; Hepatic function
MeSH Terms: conditions — Liver Diseases; Digestive System Diseases | interventions — Liver Extracts; Needles; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- liver function (Other): Subjects undergoing laparoscopic gastric surgery will be evaluated for liver function by comparing liver tissue biopsied during surgery with tissue biopsied after 60% weight loss
  Interventions: Other: liver biopsy

INTERVENTIONS:
Other: liver biopsy — Subjects undergoing laparoscopic gastric surgery will be evaluated for liver function by comparing liver tissue biopsied during surgery with tissue biopsied after 60% weight loss
  Other Names: liver; needle; biopsy

SUMMARY:
Liver disease in the morbidly obese is thought to occur due to the long-term presence of fat deposits in the liver, resulting in inflammation and scarring of the liver over time, which reduces liver function. However, many of these patients are unaware that their liver is damaged. There is currently no consensus regarding what the long-term effects of gastric bypass surgery are on pre-existing liver disease in morbidly obese patients. This study will determine the long-term effects on the liver after this type of surgical procedure.

DETAILED DESCRIPTION:
Before or on the day of surgery liver function will be determined using the DDG-2001 Analyzer. This monitor is able to detect the concentration of a dye called indocyanine green dye (ICG) when present in the blood stream. A dose of 0.5 mg/kg of ICG will be injected into an IV in the arm. Over approximately fifteen minutes the DDG-2001 Analyzer will determine how quickly the liver removes the dye ICG from the blood stream. This value represents how well the liver is functioning. Blood samples are drawn before injection of ICG to measure liver function using standard liver function tests.

This same routine for injecting ICG and obtaining blood for routine liver function tests will happen one more time, after surgery, once the subject has lost a significant amount of the original weight (60% of excess weight). This amount of weight loss typically occurs between 12 to 18 months after gastric bypass surgery. This second ICG measurement will occur during an outpatient follow-up visit to CCF.

A biopsy will be taken from the liver during surgery. A second biopsy taken after the 60% weight loss will be compared to determine the effect of this surgery on the liver.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 40.
2. Documented failed non-surgical treatment for morbid obesity.
3. Ability to undergo long-term follow-up after LGBS.

Exclusion Criteria:

1. BMI < 40.
2. Subject age < 18 years.
3. Inability to undergo long-term follow-up after LGBS (living distance > 300 miles).
4. Patients with known ESLD.
5. Patients found to have evidence of ESLD during preoperative evaluation for LGBS including portal hypertension, ascites, and coagulopathy.
6. Patients with known iodine sensitivity or allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-06; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M. Parker, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Roux-en-Y Gastric Bypass (RYGB): Before the treatment of RYGB surgery, eligible patients had preoperative liver function assessment including biochemical testing: AST, ALT, ALK, total bilirubin, albumin, and prothrombin (PT). During RYGB, a core liver biopsy was conducted. Serum lipid profiles and HbA1c values were medially optimized. Patients were asked to refrain from alcohol use for several preoperative days and discontinue hepatotoxic medications. Once patients lost 60% of their preoperative excess weight or weight loss had plateaued after RYGB surgery, they were reassessed on liver function(same as preoperative) and histology. Patients who had stable weight loss and were found to have clinically important liver damage as determined by liver biopsy at the time of RYGB were offered with repeat percutaneous ultrasound-guided liver biopsies after RYGB.
Period: Overall Study
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Started | 106
Completed | 105
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Five patients were missing on this varialbe
  Participants
    number analyzed (Participants) | 101
    Female | 70
    Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 90
  More than one race | 0
  Unknown or Not Reported | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 48 (8)
Obesity Level [Count of Participants; unit: Participants] — Morbid obesity is BMI between 35 - 40 Kg/m^2; Severe obesity is BMI greater than 40 kg/m^2.
  Participants
    Morbid Obesity | 93
    Severe Obesity | 11
    Other | 2
Duration of Obesity [Mean (Standard Deviation); unit: years] — Population: Two patients were missing on this variable
  years
    number analyzed (Participants) | 104
    (all) | 26 (12)

OUTCOME MEASURES:

1. Primary Outcome: Aspartate Transaminase (AST) Change
Description: To assess the liver function change from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure minus versus before the procedure)
Time Frame: from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure
Population: 84 patients did not have AST measured after the surgery
Measure: Mean (99.8% Confidence Interval); unit: U/L
Groups:
- Roux-en-Y Gastric Bypass (RYGB): Before the treatment of RYGB surgery, eligible patients had preoperative liver function assessment including biochemical testing: AST, ALT, ALK, total bilirubin, albumin, and prothrombin (PT). During RYGB, a core liver biopsy was conducted. Serum lipid profiles and HbA1c values were medially optimized. Patients were asked to refrain from alcohol use for several preoperative days and discontinue hepatotoxic medications.
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
U/L | -6.32 [-15.6 to 2.94]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.03, paired t-test; Mean Difference (Net) = -6.32, 99.8% CI 2-sided [-15.6 to 2.94]

2. Primary Outcome: Alanine Transaminase (ALT) Change
Description: as for outcome 1
Time Frame: as for outcome 1
Population: 84 patients did not have ALT measured
Measure: Median (99.8% Confidence Interval); unit: U/L
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
U/L | -7.56 [-22 to 6.83]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -7.56, 99.8% CI 2-sided [-22.0 to 6.83]

3. Primary Outcome: Alkaline Phosphate (ALK)
Description: To assess the liver function change from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure
Time Frame: as for outcome 1
Measure: Mean (99.8% Confidence Interval); unit: U/L
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
U/L | 5.84 [-7.55 to 19.2]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.14, paired t-test; Mean Difference (Net) = 5.84, 99.8% CI 2-sided [-7.55 to 19.2]

4. Primary Outcome: Total Bilirubin
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Only 25 patients had their postoperative measurements taken.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
mg/dl | 0.01 [-0.15 to 0.17]

5. Primary Outcome: Albumin
Description: To assess the change in liver function from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure versus before the procedure)
Time Frame: from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure minus versus before the procedure)
Population: Only 25 patients had their postoperative measurements taken.
Measure: Mean (99.8% Confidence Interval); unit: g/dL
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
g/dL | -0.2 [-0.38 to -0.02]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p < 0.001, paired t-test; Mean Difference (Net) = -0.2, 99.8% CI 2-sided [-0.38 to -0.02]

6. Primary Outcome: Prothrombin Time (PT)
Description: To assess the change in liver function from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure minus versus before the procedure)
Time Frame: as for outcome 5
Population: Only 25 patients had their measurements taken after the procedure.
Measure: Mean (99.8% Confidence Interval); unit: second
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 25
second | -0.23 [-0.68 to 0.23]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.10, paired t-test; Mean Difference (Net) = -0.23, 99.8% CI 2-sided [-0.68 to 0.23]

7. Primary Outcome: Partial Thromboplastin Time (PTT)
Description: To measure the change of PTT from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure minus versus before the procedure)
Time Frame: as for outcome 5
Population: Only 6 patients had their PTT measured after the surgery
Measure: Mean (99.8% Confidence Interval); unit: second
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 6
second | -1.72 [-8.68 to 5.25]
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.21, paired t-test; Mean Difference (Net) = -1.72, 99.8% CI 2-sided [-8.68 to 5.25]

8. Primary Outcome: Indocyanine Green (ICG) K Value
Description: To assess the liver function change from before surgery to the time when they lost 60% of their preoperative excess weight or weight loss had plateaued after this procedure (after the procedure minus versus before the procedure). ICG-k value is the slope of the decay curve of the serum ICG clearance graph, which is used to assess the liver function as it represents the rate of disappearance of ICG from blood as the liver exclusively distracts it. The lower k value means a lower rate of ICG clearance, indicating a worse liver function.
Time Frame: as for outcome 5
Population: Only 19 patients had their post-surgery ICG K measurement
Measure: Mean (99.8% Confidence Interval); unit: K(ICG) Value
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 19
K(ICG) Value | 0.01 [-0.04 to 0.06]

9. Primary Outcome: Number of Subjects of Nonalcoholic Steatohepatitis (NAS Steatosis)
Description: To compare the distribution of NAS steatosis stage from before surgery to when patients lost 60% of their preoperative excess weight or weight loss had plateaued. The NAFLD activity score (NAS) from the NASH clinical Clinic Research Network is the unweighted sum of scores for steatosis, lobular inflammation, and ballooning hepatocyte degeneration, and ranges from zero to eight points. The histological reporting for grading steatosis was based on a scale of 0 to 3, with 0 being no steatosis (<5%), 1 being mild steatosis (involving 5-33% of the biopsy specimen), 2 being moderate steatosis (involving 34-66% of the specimen), and 3 being severe (involving >66%).
Time Frame: when patients lost 60% of their preoperative excess weight or weight loss had plateaued.
Population: The outcome shows the distribution result of NAS steatosis of patients after the surgery. Only 15 people had agreed to have repeat liver biopsies.
Measure: Count of Participants; unit: Participants
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 15
Participants
  <5% | 11
  5-33% | 3
  34-66% | 1
  >66% | 0
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.002, Wilcoxon signed-rank test

10. Primary Outcome: Number of Subjects of Nonalcoholic Steatohepatitis Lobular Inflammation
Description: Lobular inflammation was similarly scored by number of foci per 200× magnification field (0 no foci: 1 < 2 foci: 2, 2-4 foci; 3, >4 foci) on biopsy specimen under microscope. This outcome was compared on its distribution before the surgery and once patients lost 60% of their preoperative excess weight or weight loss had plateaued.
Time Frame: when patients lost 60% of their preoperative excess weight or weight loss had plateaued.
Population: Only 15 people had agreed to have repeat liver biopsies.
Measure: Count of Participants; unit: Participants
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 15
Participants
  No foci | 10
  < 2 foci / 200× | 4
  2-4 foci / 200× | 1
  > 4 foci / 200× | 0
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.04, Wilcoxon signed-rank test

11. Primary Outcome: Fibrosis
Description: Fibrosis was measured from before surgery to after surgery once they lost 60% of their preoperative excess weight or weight loss had plateaued through biopsies
Time Frame: after surgery once they lost 60% of their preoperative excess weight or weight loss had plateaued
Population: Only 15 patients had repeat liver biopsies
Measure: Count of Participants; unit: Participants
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 15
Participants
  None | 6
  Perisinusoidal or periportal | 0
  1A - Mild, zone 3, perisinusoidal | 0
  1B - Moderate, zone 3, perisinusoidal | 1
  1C - Portal/periportal | 5
  2 - Perisinusoidal and portal/periportal | 2
  3 - Bridging fibrosis | 1
  4 - Cirrhosis | 0
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.005, Wilcoxon signed-rank test

12. Primary Outcome: Nonalcoholic Steatohepatitis (NAS) Hepatocyte Balloon
Description: Ballooning hepatocyte degeneration was scored as 0 (absent), 1 (few, difficult to identify), 2 (many, easily identified). This was to assess the change in the distribution of NAS hepatocyte ballon between before the surgery and once patients lost 60% of their preoperative excess weight or weight loss had plateaued
Time Frame: once patients lost 60% of their preoperative excess weight or weight loss had plateaued after surgery
Population: Only 15 patients had repeat liver biopsies
Measure: Count of Participants; unit: Participants
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 15
Participants
  Absent | 12
  Few Balloon Cells | 3
  Many cells / prominent ballooning | 0
Statistical Analysis 1: Comparison: Roux-en-Y Gastric Bypass (RYGB); Test type: Superiority; p = 0.001, Wilcoxon signed-rank test

13. Secondary Outcome: Diagnostic Accuracy-AST
Description: AST was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 101
probability | 72 [61 to 82]

14. Secondary Outcome: Diagnostic Accuracy-ALT
Description: ALT was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate and the y-axis is the true positive rate. The AUC of ROC represents the performance of diagnostic measures/models, the higher score means better performance in general. The range of AUC is from 0 to 1.0.
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 101
probability | 76 [66 to 85]

15. Secondary Outcome: Diagnostic Accuracy-ALK
Description: ALK was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate and the y-axis is the true positive rate. The AUC of ROC represents the performance of diagnostic measures/models, the higher score means better performance in general. The range of AUC is from 0 to 1.0.
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 101
probability | 65 [53 to 77]

16. Secondary Outcome: Diagnostic Accuracy-total Bilirubin
Description: The total bilirubin was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC of ROC represents the performance of diagnostic measures/models, the higher score means better performance in general. The range of AUC is from 0 to 1.0.
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 101
probability | 53 [41 to 64]

17. Secondary Outcome: Diagnostic Accuracy-PT
Description: PT was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 98
probability | 54 [41 to 67]

18. Secondary Outcome: Diagnostic Accuracy-PTT
Description: PTT (Partial Thromboplastin Time) was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 36
probability | 46 [26 to 66]

19. Secondary Outcome: Diagnostic Accuracy-ICG k Value
Description: ICG k value was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 100
probability | 53 [41 to 66]

20. Secondary Outcome: Diagnostic Accuracy-albumin
Description: Albumin was measured before RYGB surgery and was used to fit a univariate logistic model to predict clinically asymptomatic but significant fatty liver, including NASH and NASH plus fibrosis. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 99.4% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Measure: Number (99.4% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 101
probability | 55 [43 to 66]

21. Secondary Outcome: Diagnostic Accuracy-multiple Factor
Description: We also built a multivariable model using all preoperative liver function tests and ICG k clearance values to predict NASH (nonalcoholic steatohepatitis) from pre-RYGB values. AUC was used to assess the prediction performance of those multiple factors. The AUC (area under the curve) of the receiver operating characteristic curve (ROC) was calculated with a 95% confidence interval. The x-axis of ROC is the false positive rate (%) and the y-axis is the true positive rate (%). The AUC value of ROC represents the performance of diagnostic measures/models, the higher value means better performance in general. The range of AUC is from 0 to 1.0 (perfect performance).
Time Frame: before RYGB surgery
Population: Because all the pre-operative liver functions (AST, ALT, ALK, bilirubin, albumin, PT, and ICG k ) were used and 98 patients had PTT measured.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Roux-en-Y Gastric Bypass (RYGB)
Number analyzed (Participants) | 98
probability | 0.82 [0.73 to 0.90]

ADVERSE EVENTS:
Arm/Group | Liver Function
All-Cause Mortality (participants affected / at risk) | 2/106
Serious Adverse Events (participants affected / at risk) | 2/106
Other Adverse Events (participants affected / at risk) | 0/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liver Function (N=106)
Death (Cardiac disorders) | 2 (2) — death, heart attach fluid in the lungs
Bowel obstruction (Gastrointestinal disorders) | 1 (1) — Patient re hospitalized, symptoms improved
pulmonary embolism, (Blood and lymphatic system disorders) | 2 (2) — rehospitalization,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No